CLINICAL TRIAL: NCT05739721
Title: Effects of Video Conferencing on First Impressions and Attractiveness
Brief Title: ZOOM First Impressions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: DeNova Research (Other)
Responsible Party: Principal Investigator, Steven H. Dayan, Doctor of Medicine, Principal Investigator, DeNova Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZOOM-SD-2021
Record Dates: First submitted 2022-04-19; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Attractiveness; Self Esteem; First Impressions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zoom meeting (camera off) (Experimental): participants will be randomly assigned to a Zoom (San Jose, CA, USA) video conference meeting with another participant of the opposite gender
  Interventions: Behavioral: Attractiveness; Behavioral: Self-Esteem; Behavioral: Trustworthiness
- In person meeting (blindfolded) (Experimental): Once all subjects have been selected and enrolled in the study, participants will be randomly assigned for an in-person meeting.
  Interventions: Behavioral: Attractiveness; Behavioral: Self-Esteem; Behavioral: Trustworthiness
- Zoom meeting (camera on) (Experimental): participants will be randomly assigned to a Zoom (San Jose, CA, USA) video conference meeting with another participant of the opposite gender
  Interventions: Behavioral: Attractiveness; Behavioral: Self-Esteem; Behavioral: Trustworthiness
- In person meeting (no blindfold) (Experimental): Once all subjects have been selected and enrolled in the study, participants will be randomly assigned for an in-person meeting.
  Interventions: Behavioral: Attractiveness; Behavioral: Self-Esteem; Behavioral: Trustworthiness

INTERVENTIONS:
Behavioral: Attractiveness — Visual attractiveness scale 0-7
Behavioral: Self-Esteem — Self Esteem scale
Behavioral: Trustworthiness — Trustworthiness scale 0-7

SUMMARY:
Participants (random) will have a conversation with each other over zoom initially with their cameras off and then rate each other on attractiveness, first impressions, and self-esteem. Then both participants will turn their cameras back on and have another conversion and then again rate each other. The ratings are confidential and will not be shared with the other person.

Two months later the participants will come to the study clinic office and have an in-person conversation with someone new and rate each other.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of ages 21-39.
2. Subjects that understand the purpose and aspects of the study, freely sign the consent and complete the required treatment and follow up visit.
3. Subjects must all be able to speak English fluently.
4. Subjects must have access to video camera technology.
5. Fully Vaccinated against covid-19

Exclusion Criteria:

1. Participants younger than 21 or older than 40 will not be included.
2. Subjects who are pregnant or nursing.
3. Imprisoned populations.
4. Subjects who are unable to travel to the clinic.
5. Subjects that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required virtual session and follow-up visit will also be excluded.
6. Any subject that is not fully vaccinated against covid-19

Ages: 21 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 20 participants that identify as male and 20 participants that identify as female
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
First Impressions | 8 weeks
  The defined categories of first impressions include: Social skills, academic performance, dating success, occupational success, attractiveness, financial success, relationship success, and athletic success. The scale ranges from a score of 1 (less desirable) to 10 (most desirable). Scores closer to 10 signify a more positive outcome.
Trustworthiness scale | 8 weeks
  Scale 0 (disagree) - 7 (agree). Scores closer to 7 signify a more positive outcome.
Overall Attractiveness | 8 weeks
  Scale 0 (disagree) - 7 (agree). Scores closer to 7 signify a more positive outcome.

SECONDARY OUTCOMES:
Self-Esteem | 8 weeks
  The Rosenberg Self-Esteem Scale is a 10-item self-report measure of global self-esteem. It consists of 10 statements related to overall feelings of self-worth or self-acceptance. The items are answered on a four-point scale ranging from strongly agree, agree, disagree, and strongly disagree.

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States